CLINICAL TRIAL: NCT04273711
Title: Can Thyroidectomy be Considered Safe in Obese Patients? Retrospective Cohort Study
Brief Title: Can Thyroidectomy be Considered Safe in Obese Patients?
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Fabio Medas, Principal Investigator, University of Cagliari
Other Study IDs: NP20193369
Record Dates: First submitted 2020-02-13; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Thyroid; Surgery--Complications
MeSH Terms: conditions — Obesity; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patients
- Non-obese patients

SUMMARY:
Obesity is a growing public health concern in most western countries. More and more patients with high body mass index (BMI) are undergoing surgical procedures of all kinds and, in this context, obese patients are undergoing thyroid surgery more than ever before. This study showed that obesity, in the field of thyroid surgery, is not associated with any increase of postoperative complications. Thus, it is possible to conclude that thyroidectomy can be performed safely in obese patients.

DETAILED DESCRIPTION:
Background: Obesity is a growing public health concern in most western countries. More and more patients with high body mass index (BMI) are undergoing surgical procedures of all kinds and, in this context, obese patients are undergoing thyroid surgery more than ever before. The aim of the present study was to evaluate whether thyroidectomy can be considered safe in obese patients.

Methods: Patients undergoing thyroidectomy in our Unit between January 2014 and December 2018 were retrospectively analysed. Patients were divided into 2 groups: those with BMI < 30 kg/m2 were included in Group A, while those with BMI ≥ 30 kg/m2 in Group B.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to thyroidectomy in our Unit

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients submitted to thyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 813 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 1 year
  Occurrence of postoperative complications

SECONDARY OUTCOMES:
Operative time | 1 day
  Evaluation of operatives times

OTHER OUTCOMES:
Postoperative stay | up to 2 weeks
  Evaluation of postoperative stay

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Giorgio Calò, Study Director — University of Cagliari
Locations (1):
- Policlinico di Monserrato, Monserrato, CA, Italy